CLINICAL TRIAL: NCT02646839
Title: The Role of KIR-favorably Mismatched Haploidentical Transplantation and KIR-polymorphisms in Determining Outcomes of Children With ALL/AML/MDS Undergoing Allogeneic Hematopoietic Cell Transplantation
Brief Title: KIR Favorable Mismatched Haplo Transplant and KIR Polymorphism in ALL/AML/MDS Allo-HCT Children
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Michael Pulsipher (Other)
Collaborators: University of California, San Francisco (Other); Children's Hospital of Philadelphia (Other); Medical College of Wisconsin (Other); Ann & Robert H Lurie Children's Hospital of Chicago (Other); New York Medical College (Other); UCSF Benioff Children's Hospital Oakland (Other); Vanderbilt University (Other); Rady Children's Hospital, San Diego (Other)
Responsible Party: Sponsor-Investigator, Michael Pulsipher, Head of Section of Blood and Marrow Transplantation, Pediatric Transplantation & Cellular Therapy Consortium
Organization: Pediatric Transplantation & Cellular Therapy Consortium (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PBMTC ONC1401
Record Dates: First submitted 2015-12-21; First posted 2016-01-06 (Estimated); Last update posted 2025-05-04 (Actual); Status verified 2025-05

CONDITIONS: Acute Lymphoblastic Leukemia; Acute Myeloid Leukemia; Myelodysplastic Syndromes
Keywords: Acute Lymphoblastic Leukemia (ALL); Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS); KIR-Favorable; Haploidentical Transplantation; Allogeneic Hematopoietic Cell Transplantation
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myeloid, Acute; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | US Export: No

ARMS (1):
- KIR Favorable Transplant (Experimental): To assess in a multi-center setting whether the disease-free survival (DFS) at one-year post-HCT for children with high-risk ALL, AML and MDS can be improved following favorably KIR-mismatched haplo-HCT using a graft ex vivo depleted of T cell receptor (TCR) αβ+CD3+/CD19+ cells from CliniMacs TCR alpha-beta-Biotin system
  Interventions: Device: CliniMacs TCR alpha-beta-Biotin system

INTERVENTIONS:
Device: CliniMacs TCR alpha-beta-Biotin system — Graft ex vivo depleted of T cell receptor (TCR) αβ+CD3+/CD19+ cells

SUMMARY:
This is a phase II, open-label, non-randomized, prospective study of haploidentical transplantation using KIR-favorable donors for children with acute lymphoblastic leukemia (ALL), acute myeloid leukemia (AML) and myelodysplastic syndrome (MDS) undergoing allogeneic hematopoietic cell transplantation (HCT). The relationship of KIR2DL1 polymorphisms to survival in children with these diseases undergoing any approach to allogeneic HCT during the study time frame will also be determined.

DETAILED DESCRIPTION:
Allogeneic hematopoietic stem cell transplantation (HCT) using matched related and unrelated donors is well-accepted therapy for children with subtypes of high-risk acute lymphoblastic leukemia (ALL) and acute myeloid leukemia (AML). For the 40-50% of children who do not have matched donors available, HCT approaches have varied by center and regional preferences. HCT physicians in France and North America tend to use human leukocyte antigen (HLA)-mismatched umbilical cord blood (UCB), while those in many large centers in Germany, parts of Asia, and selected US centers favor HLA-haploidentical donors. Both approaches have improved significantly through the years for a variety of reasons, including better supportive care, cell processing techniques that now deliver more consistently high-quality products, understanding of the importance of cell dose, and key modifications of preparative and immunosuppressive regimens.

Both stem cell sources offer distinct advantages and disadvantages. T-cell-depleted haploidentical approaches with killer-cell immunoglobulin-like receptor (KIR) mismatches have been shown to lead to less relapse in patients with AML13 and, in some studies, children with ALL as well. Disadvantages to this approach have been vulnerability to viral infection and the requirement for an ex vivo T-cell depletion procedure that is currently under IND. Cord blood is readily available and is permissive of some degree of HLA mismatch, but current studies show no advantage in survival compared with matched unrelated donors. Recently, a randomized study of one vs. two UCB units based on a hypothesis of decreased relapse incidence with two units resulted in equivalent outcomes in both arms. Neutrophil engraftment and immune recovery after UCB transplantation is relatively slow, leading to a higher risk of transplant-related mortality; in addition, larger patients require two cord units, dramatically increasing the cost of stem cell procurement. No direct comparisons of these two stem cell sources (haploidentical vs. UCB) have been performed in pediatric patients.

Recently, investigators at St. Jude Children's Research Hospital published excellent outcomes using haploidentical donors with grafts depleted for CD3+ cells by an ex vivo Miltenyi CliniMACS system. Their recent cohort of AML and ALL patients treated without total body irradiation (TBI) had a 5-year survival of 88±15% in 19 consecutive patients, with 17 surviving long-term and disease-free and only 2 patients died of progressive leukemia. These results compared favorably with the 5-year survival of 70±38% for transplantations using matched siblings and 61±17% for matched unrelated donors treated with identical leukemia protocols with indications for transplantation defined a priori. These preliminary results suggest that a strategy of using favorable KIR-mismatched haploidentical transplantation may lead to a better outcome than other alternative donor approaches without the side effects of TBI. This protocol is a phase II trial seeking to establish the feasibility and preliminary outcomes with this approach in a multi-institutional setting.

In addition to KIR-HLA matching, KIR allele polymorphism may also affect transplant outcomes.Recent data from St. Jude showed that in 312 pediatric HCTs, the patients who received a donor graft containing the functionally stronger KIR2DL1 allele with arginine at amino acid position 245 (KIR2DL1-R245) had better survival (p=0.0028) and a lower relapse rate (p=0.022) than those who received a donor graft that contained only the functionally weaker KIR2DL1 allele with cysteine at the same position (KIR2DL1-C245). Patients who received a KIR2DL1-R245-positive graft with an HLA-C receptor-ligand mismatch had the best survival (p=0.00004) and lowest risk of leukemia relapse (p=0.005). Thus, both KIR-HLA matching and KIR allele polymorphism have prognostic value. We will attempt to prospectively confirm these results in this multicenter trial.

ELIGIBILITY:
Inclusion Criteria:

2.3.1 Inclusion Criteria for the Biology (KIR2DL1 Polymorphisms/ALL MRD), Comparative Outcomes, and Cost Effectiveness Trial

1. Any patient with ALL, AML, or MDS who is deemed eligible for and undergoes HCT at participating centers who provides consent for the KIR2DL1 polymorphisms, comparative outcomes and cost-effectiveness portion of the trial.
2. Any ALL patient undergoing allogeneic HCT at participating centers is eligible for the ALL deep sequence MRD portion of the trial.
3. Patients ineligible for the KIR-favorable haploidentical phase II trial who require T-cell depletion may be treated using TCR αβ+CD3+/CD19+ cell depletion. These patients will be followed descriptively on this portion of the trial. Preparative regimen will be at the discretion of the transplant center, but the options associated with this protocol are recommended.

2.3.2 Inclusion Criteria for the KIR-favorable Haploidentical Phase II trial:

1. Age < 22 years
2. Disease and disease status:

   * ALL high-risk in first remission (<5% blasts by morphology pre-transplant) meeting criteria for transplant. Example CR1 indications: induction failure (>5% blasts by morphology on post-induction BM), minimal residual disease greater than or equal to 1% marrow blasts by morphology after induction, minimal residual disease by flow cytometry >0.01% after consolidation, hypodiploidy (<44 chromosomes), persistent or recurrent cytogenetic or molecular evidence of disease during therapy requiring additional therapy after induction to achieve remission (e.g. persistent molecular BCR-ABL positivity).
   * ALL in second remission: B-cell; early (less than or equal to 36 months from initiation of therapy) BM relapse, late BM relapse with MRD >0.1% by flow cytometry after first induction therapy; T-cell or Ph+ with BM relapse at any time; very early (less than 18 months from initiation of therapy) isolated extramedullary relapse (T or B-cell)
   * Myelodysplastic syndrome (MDS): Any 2001 WHO classification subtype (Appendix I). RAEB-2 patients may proceed directly to transplant, but may also receive induction chemotherapy before transplant. Patients with ≥20% morphologic marrow blasts will require induction therapy to reduce morphologic marrow blasts below 5% before transplant.
   * High-risk AML defined as monosomy 5, del 5q, monosomy 7, M6, M7, t(6;9), FLT3-ITD, or patients who have greater than or equal to 25% blasts by morphology after induction, or who do not achieve CR after 2 courses of therapy. Also, patients with ≥ 0.1% MRD or evidence of progressive extramedullary disease after induction chemotherapy.
   * AML in second or subsequent morphologic remission.
3. Has not received a prior allogeneic hematopoietic stem cell transplant.
4. Does not have a suitable HLA-matched sibling donor available for stem cell donation.
5. Does not have a suitable matched or single antigen mismatched related or unrelated donor available at any time (noted by search), or it is in the patient's best interest as judged by the attending to move forward with stem cell transplantation rather than wait for an unrelated donor to become available (refer to subsection 2.5.1 for further details).
6. Has a suitable HLA KIR favorable haploidentical matched family member available for stem cell donation.
7. Karnofsky Index or Lansky Play-Performance Scale ≥ 60 % on pre-transplant evaluation. Karnofsky scores must be used for patients > 16 years of age and Lansky scores for patients < 16 years of age.
8. Able to give informed consent if > 18 years, or with a legal guardian capable of giving informed consent if < 18 years.
9. Adequate organ function (within 4 weeks of initiation of preparative regimen), defined as:

   * Pulmonary: FEV1, FVC, and corrected DLCO must all be ≥ 50% of predicted by pulmonary function tests (PFTs). For children who are unable to perform for PFTs due to age, the criteria are: no evidence of dyspnea at rest and no need for supplemental oxygen.
   * Renal: Creatinine clearance or radioisotope GFR ³ 70 mL/min/1.73 m2 or a serum creatinine based on age/gender as follows:

Age Maximum Serum Creatinine (mg/dL) Male Female 1 to < 2 years 0.6 0.6 2 to < 6 years 0.8 0.8 6 to < 10 years 1 1 10 to < 13 years 1.2 1.2 13 to < 16 years 1.5 1.4

≥ 16 years 1.7 1.4 The threshold creatinine values in this Table were derived from the Schwartz formula for estimating GFR utilizing child length and stature data published by the CDC.45

* Cardiac: Shortening fraction of ≥ 27% by echocardiogram or radionuclide scan (MUGA) or ejection fraction of ≥ 50% by echocardiogram or radionuclide scan (MUGA), choice of test according to local standard of care.
* Hepatic: \SGOT (AST) or SGPT (ALT) < 5 x upper limit of normal (ULN) for age. Conjugated bilirubin < 2.5 mg/dL, unless attributable to Gilbert's Syndrome.

Exclusion Criteria:

1. Pregnant or lactating females are ineligible as many of the medications used in this protocol could be harmful to unborn children and infants.
2. Patients with HIV or uncontrolled fungal, bacterial or viral infections are excluded. Patients with history of fungal disease during induction therapy may proceed if they have a significant response to antifungal therapy with no or minimal evidence of disease remaining by CT evaluation.
3. Patients with active CNS leukemia or any other active site of extramedullary disease at the time of enrollment are not permitted. Note: Those with prior history of CNS or extramedullary disease, but with no active disease at the time of pre-transplant workup, are eligible.
4. Patients with genetic disorders (generally marrow failure syndromes) prone to secondary AML/ALL with known poor outcome are not eligible (Fanconi Anemia, Kostmann Syndrome, Dyskeratosis Congenita, etc).

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-10; Primary Completion 2025-11 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival at 1 year post HCT | 1 year
1 yr disease free survival of patients transplanted with donors homozygous for KIR2DL1-C245 will be compared to patients with donors hetero- or homozygous for KIRD2DL1-R245 polymorphisms | 1 year

SECONDARY OUTCOMES:
1- and 2-year overall survival (OS) for children undergoing TCR αβ+CD3+/CD19+ cell depleted favorably KIR-mismatched haplo-HCT | 2 years
Cumulative incidence of neutrophil and platelet engraftment, primary and secondary rejection, NTM, and relapse in KIR favorable haplo-HCT recipients | 1 year
Cumulative incidence of overall grades II-IV and III-IV acute GVHD in KIR favorable haplo-HCT recipients | 5 years
Compare the 2-year DFS and OS of patients transplanted using favorably KIR-mismatched haplo-HCT with other ALL, AML, and MDS patients concurrently transplanted using other approaches at the participating centers. | 1 year
Compare the 2-year DFS and OS of patients transplanted using favorably KIR-mismatched haplo-HCT with other ALL, AML, and MDS patients concurrently transplanted using 4/6 and 5/6 HLA-matched cord blood reported to the CIBMTR | 1 year
Test sensitivity of flow cytometry MRD for all patients; in ALL patients, compare flow cytometry MRD with IgH and TCR next-generation-sequencing (NGS) MRD pre- and post-HCT for predicting relapse, DFS, and OS in children undergoing allog-HCT. | 1 year
To compare costs of transplantation using favorably KIR-mismatched haplo-HCT with patients receiving alternative donor transplantation at centers participating in the trial | 1 year
1- and 2-year event free survival (DFS) for children undergoing TCR αβ+CD3+/CD19+ cell depleted favorably KIR-mismatched haplo-HCT | 2 years
Cumulative incidence of chronic GVHD in KIR favorable haplo-HCT recipients. | 1 year
Cumulative incidence of mild, moderate, and severe cGVHD | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Pulsipher, MD, Principal Investigator — Children's Hospital Los Angeles
Locations (11):
- United States (11):
  - Children's Hospital Los Angeles, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - Stanford University Medical Center, Palo Alto, California
  - Rady Children's Hospital, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Lurie Children's Hospital, Chicago, Illinois
  - New York Medical Center, Valhalla, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Vanderbilt University - Monroe Carell Jr. Children's Hospital, Nashville, Tennessee
  - University of Utah, Primary Children's Hospital, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dvorak CC, Long-Boyle JR, Holbrook-Brown L, Abdel-Azim H, Bertaina A, Vatsayan A, Talano JA, Bunin N, Anderson E, Flower A, Lalefar N, Higham CS, Kapoor N, Klein O, Odinakachukwu MC, Cho S, Jacobsohn DA, Collier W, Pulsipher MA. Effect of rabbit ATG PK on outcomes after TCR-alphabeta/CD19-depleted pediatric haploidentical HCT for hematologic malignancy. Blood Adv. 2024 Dec 10;8(23):6003-6014. doi: 10.1182/bloodadvances.2024012670. PMID 39042892
- [Derived] Pulsipher MA, Ahn KW, Bunin NJ, Lalefar N, Anderson E, Flower A, Cairo MS, Talano JA, Chaudhury S, Kitko CL, Duke JL, Monos D, Leung W, Dvorak CC, Abdel-Azim H. KIR-favorable TCR-alphabeta/CD19-depleted haploidentical HCT in children with ALL/AML/MDS: primary analysis of the PTCTC ONC1401 trial. Blood. 2022 Dec 15;140(24):2556-2572. doi: 10.1182/blood.2022015959. PMID 35776909